CLINICAL TRIAL: NCT05803720
Title: Development of an Online Provider Intervention to Address Intersectional Stigma and Medical Mistrust in People Living With HIV
Brief Title: HIV Provider Intervention to Address Intersectional Stigma and Medical Mistrust
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: California Prevention Training Center (Unknown); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lu Dong, Full Behavioral/Social Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-N0035
Record Dates: First submitted 2023-02-14; First posted 2023-04-07 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stigma, Social
MeSH Terms: conditions — Social Stigma | interventions — Seroconversion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the study condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider Intervention (Experimental): The intervention will consist of psychoeducation and skills-building for HIV care providers to gain the knowledge and skills needed to address intersectional stigma and medical mistrust with patients. The intervention will be online and conducted in groups.
  Interventions: Behavioral: Provider Intervention on Addressing Intersectional Stigma and Medical Mistrust in Patients with HIV
- Control (No Intervention): No intervention control

INTERVENTIONS:
Behavioral: Provider Intervention on Addressing Intersectional Stigma and Medical Mistrust in Patients with HIV — The intervention will consist of psychoeducation and skills-building for HIV care providers to gain knowledge and skills needed to address intersectional stigma and medical mistrust with patients. The intervention will be online and conducted in groups.
  Arms: Provider Intervention

SUMMARY:
Intersectional stigma and medical mistrust are prevalent among Black and Latina/Latino Americans living with HIV and are key contributors to racial/ethnic health disparities; yet, there are no evidence-based provider-level interventions available for HIV care providers to address intersectional stigma and medical mistrust with patients. The investigators propose to develop an online provider intervention, with community stakeholders' input, that provides psychoeducation and skills-building around addressing intersectional stigma and medical mistrust with patients. The investigators will conduct a pilot randomized controlled trial with 60 HIV care physicians (30/condition) to test the acceptability and feasibility of the online intervention and to determine preliminary effects (against a no-intervention control group) on providers' use of skills and HIV care delivery outcomes at baseline, immediate post, and 6-month follow-up.

DETAILED DESCRIPTION:
The first aim will be an intervention development process that involves engaging community stakeholders to incorporate their input on the intervention manual and working with a provider training organization to develop an online platform for the initial pilot testing. The intervention will include psychoeducation and skills-building for providers to address intersectional stigma and mistrust, tailored to HIV care. This aim will include a usability test of the online intervention in 10 HIV clinical care providers. The second aim will be to conduct a pilot randomized controlled trial to compare two conditions (i.e., online provider intervention versus no-intervention control) on provider training outcomes (e.g., providers' use of skills learned in the intervention) and HIV care delivery outcomes (e.g., the estimated percentage of patients lost to care in the past year) measured at baseline, immediate post-intervention, and 6-month follow-up. Clinical providers (N = 60) providing care for patients living with HIV will be randomly assigned to the online provider intervention (n = 30) or control with no intervention (n = 30). The intervention will be delivered in groups (5-10 providers per group). A mixed-methods process evaluation at immediate post-intervention will determine the acceptability, feasibility, and appropriateness of the intervention, and will be used to refine the intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical providers (including physicians, physician assistants, nurse practitioners, registered nurses/case managers) caring for patients living with HIV,
* the majority of their patients are from racial/ethnic and sexual minority groups,
* can make the time commitment to participate in the study.

Exclusion Criteria:

* not HIV clinical providers
* cannot make the time commitment to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lu Dong, PhD, Principal Investigator — RAND
Locations (1):
- RAND Corporation, Santa Monica, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Provider Training Group: Providers in the training intervention group participated in a multi-component educational program designed to improve communication with patients experiencing intersectional stigma and medical mistrust in HIV care. The training included three parts: (1) a 30-40 minute pre-recorded video introducing key concepts, supported by patient narratives and research evidence; (2) a 60-minute live virtual session led by faculty from the California Prevention Training Center, featuring interactive discussion and role-play exercises to practice communication strategies; and (3) a downloadable self-paced workbook with case scenarios and reflection prompts. The intervention aimed to build provider skills in recognizing and addressing patient mistrust and stigma using respectful, autonomy-supportive communication techniques. Participants completed assessments at baseline, immediately post-training, and at 6-month follow-up.
- No Training Control Group: Providers in the control group did not receive any training during the study period. They completed study assessments at baseline, immediately post-intervention (parallel to the intervention group's timeline), and at 6-month follow-up. After study completion, they were offered access to the training materials for ethical and educational purposes.
Period: Overall Study
Arm/Group | Provider Training Group | No Training Control Group
Started | 29 | 30
Received the allocated intervention | 27 | 28
Completed post assessment | 25 | 23
Completed 6-month assessment | 25 | 25 (Two individuals are lost for the control group at 6-month (n=2). One individual is lost due to the loss of contact. Three individuals who are lost to follow up at Post but participated in the 6-month follow-up.)
Completed | 25 | 25
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Family leave/emergency | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Provider Training Group: Participants received a three-part training on addressing medical mistrust and intersectional stigma in HIV care. The training included a 1-hour recorded module, a 2-hour live role-play session, and a self-paced workbook. Content focused on using validation and motivational interviewing strategies to improve provider communication.
- Control Group: Participants in the control group did not receive any training during the study period. They completed the same baseline, post, and follow-up assessments as the intervention group for comparison purposes.
- Total: Total of all reporting groups
Arm/Group | Provider Training Group | Control Group | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants in the control condition did not complete demographic information (i.e., missing data on age)
  years
    number analyzed (Participants) | 29 | 28 | 57
    (all) | 42.4 (13.72) | 42.82 (10.58) | 42.61 (12.17)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: 2 participants in the control condition did not complete demographic information (i.e., missing data on gender identification)
  Participants
    Male: number analyzed (Participants) | 29 | 28 | 57
    Male | 8 | 8 | 16
    Female: number analyzed (Participants) | 29 | 28 | 57
    Female | 18 | 17 | 35
    Man, Female-to-Man (FTM): number analyzed (Participants) | 29 | 28 | 57
    Man, Female-to-Man (FTM) | 1 | 2 | 3
    Prefer not to answer: number analyzed (Participants) | 29 | 28 | 57
    Prefer not to answer | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Training group: 1 identified as Man (female to man, 2 prefer not to answer Control group: 2 identifies as Man (female to man), 1 prefer not to answer, also 2 missing this variable in baseline survey.
  Participants
    number analyzed (Participants) | 26 | 25 | 51
    Female | 18 | 17 | 35
    Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 26 | 23 | 49
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 16 | 13 | 29
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Helpful/Empathetic Responses Toward Medial Mistrust in Hypothetical Patient Scenarios
Description: Helpful/empathic responses will be operationalized as the number of motivational interviewing (MI)-consistent statements and validation used in the written responses; this variable will be obtained by coding the responses to the Helpful Response Questionnaire using the Motivational Interviewing Skills Coding for the number of validation and MI-consistent statements used in the written response. This measure is a count variable and the values ranging above or equal to 0 (no maximum). Higher values represent a better outcome.
Time Frame: Baseline, 2-monts after the baseline assessment, and 6-month follow-up
Population: Participants dropped out or cannot be reached after baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Training Group | Control Group
Number analyzed (Participants) | 29 | 30
score on a scale
  Baseline | 9.81 (2.60) | 9.26 (1.75)
  2-month after the baseline assessment: number analyzed (Participants) | 25 | 23
  2-month after the baseline assessment | 10.68 (3.99) | 8.90 (2.05)
  6-month follow-up: number analyzed (Participants) | 25 | 25
  6-month follow-up | 9.29 (2.94) | 9.16 (2.13)

2. Primary Outcome: Provider Use of Strategies Learned in the Provider Intervention in a Role-play Simulation of Hypothetical Patient Scenarios
Description: Provider use of strategies learned in the provider intervention in a role-play simulation will be obtained through coding that will be developed specifically for this study based on existing coding schemes (e.g., Motivational Interviewing Skills Coding, as appropriate). This variable will be calculated as the total number of training-consistent strategies used during the role-play simulation. This measure is a count variable and the values ranging above or equal to 0 (no maximum). Higher values represent a better outcome.
Time Frame: Baseline and 2-month after the baseline assessment
Population: Participants dropped out or cannot be reached after baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Training Group | Control Group
Number analyzed (Participants) | 29 | 30
score on a scale
  Training-consistent codes at Baseline | 8.04 (2.96) | 7.94 (2.37)
  Training-consistent codes at Post (2 months after baseline assessment): number analyzed (Participants) | 25 | 23
  Training-consistent codes at Post (2 months after baseline assessment) | 8.60 (3.07) | 7.56 (2.30)

3. Primary Outcome: Provider Use of Strategies Learned in the Provider Intervention in a Role-play Simulation of Hypothetical Patient Scenarios
Description: Provider use of strategies learned in the provider intervention in a role-play simulation will be obtained through coding that will be developed specifically for this study based on existing coding schemes (e.g., Motivational Interviewing Skills Coding, as appropriate). This variable will be calculated as the total number of training-inconsistent strategies used during the role-play simulation. This measure is a count variable and the values ranging above or equal to 0 (no maximum). Higher values represent a better outcome.
Time Frame: Baseline and 2-month after the baseline assessment
Population: Participants dropped out or cannot be reached after baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Provider Training Group | Control Group
Number analyzed (Participants) | 29 | 30
score on a scale
  Training-inconsistent codes at Baseline | 0.33 (0.54) | 0.67 (0.78)
  Training-inconsistent codes at Post (2 months after baseline assessment): number analyzed (Participants) | 25 | 23
  Training-inconsistent codes at Post (2 months after baseline assessment) | 0.29 (0.51) | 0.53 (0.47)

ADVERSE EVENTS:
Time Frame: Approximately 6 months during study participation
Description: None reported
Arm/Group | Provider Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

LIMITATIONS AND CAVEATS:
The study sample consisted of self-selected HIV providers, which may limit the generalizability of findings to broader provider populations. The study used role-play simulations which were limited in capturing provider interaction with patients in real-world clinical encounters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT05803720/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05803720/ICF_000.pdf